CLINICAL TRIAL: NCT06270459
Title: Telerehabilitation Robotics for Upper Limb Rehabilitation After STroke (TRUST): a Study of Multi-cluster Adoption
Brief Title: Telerehabilitation Robotics for Upper Limb Rehabilitation After STroke
Acronym: TRUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2023/00954
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study is a multi-site prospective clinical trial, with single-arm study design with independent assessment of outcome measures (i.e., robotic metrics, standardized outcomes, quality of life, subjective measures).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HMAN robot @ Home (Experimental): 4 weeks of daily HMAN robot training at participant's home (for up to 120 minutes per day with rest breaks) interspersed with 2 sessions of conventional therapy sessions (COTS) and 2 additional COTS upon completion of 4-week HMAN robot training at home.
  Interventions: Device: HMAN Robot

INTERVENTIONS:
Device: HMAN Robot — The HMAN is certified as a CE class 2A upper limb rehabilitation robot suitable for hospital, clinic and home-based use in 2020 by Health Sciences Authority, Singapore. It has since been employed in post-stroke neurorehabilitation therapy and assessment of sensorimotor functions in stroke patients.

SUMMARY:
There has been an observed decrease in motor and functional ability and non-use of the impaired limb in chronic patients. This is due to the immediate drop in intensive daily therapy (5 days per week for 3 hours/day) that is usually provided during the inpatient (acute) phase upon discharge from the hospital.

In this study, the investigators plan to address the low dosage of therapy in the post-acute discharge phase for stroke survivors.

DETAILED DESCRIPTION:
Current models of care in public healthcare institutions (PHI) cannot provide daily or frequent access to RAT without increasing burden and expenditure in direct healthcare resources. Shifting from the existing hospital-based model of care towards a home-centered model based deploying portable RAT, would ensure that patients can continue to receive intensive therapy after discharge and during the chronic phase of stroke.

More recently, RAT deploying table-top, portable, less complex, upper limb end effectors enable clinic-to-home transitions may offer decentralized therapy, minimally supervised by therapists as a potential means to bridge various gaps in access to RAT such as scheduling, physical or social barriers, distances and hospital lockdowns related to viral pandemics.

This study aims to explore the utilization, feasibility and acceptability using a multi-cluster deployment and adoption of a decentralised robot-aided telerehabilitation (RATR) clinical programme supported by AI-enabled platform, with remote monitoring by clinic therapists

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stroke (ischaemic or haemorrhagic) confirmed by admitting doctors and CT, CT angiography or MRI brain imaging.
2. Age 21 to 90 years, both males and females.
3. At least > 28 days post stroke.
4. Upper limb motor impairment of Fugl-Myer Motor Assessment (FMA) scale 10 to 60
5. Has a stable home abode and a carer/ NOK to supervise home based exercise.
6. Ability to sit supported continuously for 60 minutes.
7. Montreal Cognitive Assessment (MOCA) score > 21/30
8. Able to understand purpose of research and give consent.

Exclusion Criteria:

1. Non-stroke related causes of arm motor impairment.
2. Medical conditions incompatible with research participation: uncontrolled medical illnesses (hypertension or diabetes, ischaemic heart disease, congestive heart failure, bronchial asthma, end stage renal/liver/heart/lung failure, unresolved cancers.
3. Anticipated life expectancy of < 6 months.
4. Inability to tolerate sitting continuously for 60 minutes.
5. Local factors potentially worsened by intensive robot-aided arm therapy and computer-based training: active seizures within 3 months, spasticity of Modified Ashworth Scale grades >2 skin wounds, shoulder, arm pain VAS > 5/10, active upper limb fractures, arthritis, fixed upper limb flexion contractures.
6. Hemianesthesia of affected limb.
7. History of dementia, severe depression, agitation, or behavioural problems.
8. Pregnancy or lactation in females
9. Absence of reliable carer to provide supervision during home training

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
Compliance Rates | Through study's data collection period, up to 2 years
  Using cloud data from vendor, time (min/hours) of HMAN robot usage

SECONDARY OUTCOMES:
Fugl Meyer Motor Assessment (FMA) | Weeks 0 (baseline), Week 6 (end of HMAN @ Home), Week 8 (end of treatment phase), Week 12 (1st Follow-up), Week 24 (Last follow-up)
  Change in Fugl Meyer Motor Assessment score in the affected arm
Action Research Arm Test (ARAT) | Weeks 0 (baseline), Week 6 (end of HMAN @ Home), Week 8 (end of treatment phase), Week 12 (1st Follow-up), Week 24 (Last follow-up)
  Functional and dexterity score for upper extremities, minimum 0, maximum 57; with higher score indicating better function
Grip strength (KgF) measured by Digital Dynamometer (mean of 3 readings will be recorded) | Weeks 0 (baseline), Week 6 (end of HMAN @ Home), Week 8 (end of treatment phase), Week 12 (1st Follow-up), Week 24 (Last follow-up)
  Measured by Digital Dynamometer (mean of 3 readings will be recorded)
System Usability Scale (SUS) | Week 6 (end of HMAN @ Home)
  For evaluation of the HMAN robot's perceived usability, scaled from 1 (Strongly disagree) to 5 (Strongly Agree)
Intrinsic Motivation Inventory (IMI) | Week 6 (end of HMAN @ Home)
  To assess participants' subjective experience on usage of the HMAN robot using 4 separate subscales (Interest/Enjoyment, Perceived competence, Perceived choice, Pressure/Tension)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chua, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No